CLINICAL TRIAL: NCT06126081
Title: Clinical Efficacy of Early Left Bundle Branch Pacing for Cardiac Resynchronization Therapy Compared With Guideline-directed Medical Therapy in Heart Failure With Mild-reduced Ejection Fraction.
Brief Title: Clinical Efficacy of Early Left Bundle Branch Pacing for Cardiac Resynchronization Therapy
Acronym: Early-RESYNC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fu Wai Hospital, Beijing, China (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xiaohan Fan, Professor, MD, PhD, Fu Wai Hospital, Beijing, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1996
Record Dates: First submitted 2023-09-05; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure; Left Bundle Branch Pacing
Keywords: Heart Failure; Left Bundle Branch Pacing; Guideline-Directed Medical Therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: 1:1 randomized to two groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LBBP+GDMT group (Experimental): Patients in the LBBP+GDMT group will receive LBBP using dual-chamber device as priority and guideline-directed medical therapy. The pacing lead will be implanted at the left bundle branch and whether LBB is captured will be judged during the procedure. For patients who LBBP is failed, CRTP using triple-chamber device or LVSP by using dual-chamber device will be an alternative option according to the co-determination after consultation between doctors and patients .
  Interventions: Device: LBBP+GDMT
- GDMT group (Active Comparator): Patients in the GDMT group will receive guideline-directed medical therapy according to their complications, heart rate, blood pressure and so on. During follow-up of 6 months, patients may transfer to LBBP group if the LVEF decreased to <35% and patients accepted the device implantation.
  Interventions: Drug: GDMT

INTERVENTIONS:
Device: LBBP+GDMT — LBBP is a procedure that the pacing lead is placed at the left bundle branch to achieve electrical and mechanical synchronization by pacing the left bundle branch area with stable pacing parameters.
  Other Names: Early Resynchc
  Arms: LBBP+GDMT group
Drug: GDMT — GDMT is defined as the drug strategy for treatment of heart failure according to the current guidelines.
  Other Names: Conventional treatment
  Arms: GDMT group

SUMMARY:
This is a two-center, prospective randomized controlled trial. The aim of this study is to compare the clinical efficacy of early left bundle branch pacing for cardiac resynchronization therapy and guideline-directed medical therapy in heart failure with mild-reduced ejection fraction.

DETAILED DESCRIPTION:
Early-resync is a two-center, prospective randomized controlled trial that is designed to determine whether early left bundle branch pacing has a better impact on LV function improvement as compared with traditional guideline-directed medical therapy in heart failure with mild-reduced ejection fraction（36%≤LVEF≤50%） and complete left bundle branch block (CLBBB). Patients with symptomatic heart failure,36%≤LVEF≤50%, NYHA function class II-IV, and CLBBB（according to STRAUSS criteria) will be 1:1 randomized to LBBP+GDMT or GDMT group after enrollment and be followed at 3 and 6 months after randomization. LBBP will be performed by a double-chamber device in LBBP+GDMT group. All patients will receive GDMT. The primary endpoint is the change in the LVEF at 6 months after randomization from baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. symptomatic heart failure despite guideline-directed medical therapy for at least 3 months, NYHA class II-IV, with an EF between 35% and 50%;
3. complete LBBB meeting Strauss's standard definition
4. Signed informed consent.

Exclusion Criteria:

1. Expected survival less than 24 months;
2. Indicated for ICD or pacing therapy;
3. History of VT, VF, or hemodynamic instability;
4. History of mechanical tricuspid valve replacement;
5. Ischemic cardiomyopathy scheduled for CABG and PCI within 3 months;
6. Severe structural heart disease may necessitate cardiac surgery or heart transplantation within 1 year;
7. Pregnancy or planning for pregnancy;
8. Hypertrophic cardiomyopathy or those underwent ventricular septal defect repair, in whom the success of LBBP is anticipated to be challenging;
9. Severe renal dysfunction (eGFR < 15ml/min*1.73m^2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
ΔLVEF between baseline and 6-month follow-up | 6 months
  ΔLVEF：change in LVEF in percentage (%) between baseline and 6-month follow-up

SECONDARY OUTCOMES:
ΔLVEDD and ΔLVESV between baseline and 6-month follow-up | 6 months
  ΔLVEDD：change in LVEDD in millimeters between baseline and 6-month follow-up between two groups.
  ΔLVESV：change in LVESV in milliliters between baseline and 6-month follow-up between two groups.
The echocardiographic response rate of LVEF ≥50% | 6 months
  the percentage of patients with LVEF ≥50% at 6 month follow-up
The changes of NYHA function class between baseline and 6-month follow-up. | 6 months
  NYHA function class (from I to IV) is evaluated by clinicians at each outpatient follow-up visit;
Composite incidence rate of all-cause mortality and/or hospitalization for heart failure | 6 months
  All-cause death: including cardiovascular and non-cardiovascular deaths. Hospitalization for heart failure: an unplanned outpatient or emergency department visit or inpatient hospitalization in which the patient presented with signs and symptoms consistent with heart failure and required medication therapy.
The rate of LVEF <=35% at six-month | 6 months
  The percentage of patients with LVEF <=35% at 6 month follow-up
The changes of NT-proBNP between baseline and 6-month follow-up. | 6 months
  NT-proBNP in pg/ml was measured by performing a blood test;
The changes of 6MWD between baseline and 6-month follow-up. | 6 months
  6MWD in meters stands for "6-Minute Walk Distance." It is a common test used to assess a person's functional exercise capacity and cardiovascular endurance. During the test, the patient is asked to walk as far as possible within a span of 6 minutes in a straight path or designated walking course;
The changes of QoL between baseline and 6-month follow-up. | 6 months
  QoL stands for "Quality of Life", which is measured by The Minnesota Living with Heart Failure Questionnaire (MLHFQ). The MLHFQ is a self-administered disease-specific questionnaire for patients with HF, comprising 21 items from 0 (none) to 5 (very much). It provides a total score (range 0-105, from best to worst HRQoL).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohan Fan, PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (2):
- China (2):
  - Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The first affiliated hospital of Nanjing medical university, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No